CLINICAL TRIAL: NCT01558648
Title: Quality of Life Outcomes Following Minimally Invasive and Open Esophagectomy for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-003
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-04

CONDITIONS: Esophageal Cancer
Keywords: Minimally Invasive Esophagectomy; Open Esophagectomy; Quality of Life; 12-003
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pts having Minimally Invasive esophagectomy: This is a prospective non-randomized study comprising two surgical cohorts of esophageal cancer patients. Patients will be assigned to each of the two intervention groups, MIE versus OE, based on a combination of patient referral patterns, patient preference, and surgeon preference/expertise.
  Interventions: Behavioral: Quality of Life instruments, FACT-E, Symptom Assessment Scale, Brief Pain Inventory and Daily Analgesic Log
- Pts having open esophagectomy: This is a prospective non-randomized study comprising two surgical cohorts of esophageal cancer patients. Patients will be assigned to each of the two intervention groups, MIE versus OE, based on a combination of patient referral patterns, patient preference, and surgeon preference/expertise.
  Interventions: Behavioral: Quality of Life instruments, FACT-E, Symptom Assessment Scale, Brief Pain Inventory and Daily Analgesic Log

INTERVENTIONS:
Behavioral: Quality of Life instruments, FACT-E, Symptom Assessment Scale, Brief Pain Inventory and Daily Analgesic Log — Initial pre-operative assessment post-operative assessment in-hospital assessment at first post-operative visit (clinic visits, or by telephone or mail) assessments at 4, 8, 12, 18, and 24 months post-operatively (+/- 2 month window). For patients who have their surgery delayed, they may be asked to complete another, more updated set of pre-surgery surveys. For the dysphagia score and CT Scan vs EUS subset will be a dysphagia questionnaire, administered at the time of the initial clinic visit.
  Groups: Pts having Minimally Invasive esophagectomy
Behavioral: Quality of Life instruments, FACT-E, Symptom Assessment Scale, Brief Pain Inventory and Daily Analgesic Log — Initial pre-operative assessment post-operative assessment in-hospital assessment at first post-operative visit (clinic visits, or by telephone or mail) assessments at 4, 8, 12, 18, and 24 months post-operatively (+/- 2 month window). For patients who have their surgery delayed, they may be asked to complete another, more updated set of pre-surgery surveys. For the dysphagia score and CT Scan vs EUS subset will be a dysphagia questionnaire, administered at the time of the initial clinic visit.
  Groups: Pts having open esophagectomy

SUMMARY:
The goal of this study is to evaluate how surgery for esophageal cancer affects the patient's quality of life over time. The investigators hope this study will provide important information that can be used to improve the quality of life of patients with esophageal cancer. This study will also look at how standard tests and information collected from the patients difficulty swallowing can predict the extent of their esophageal cancer before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of esophageal cancer, stages I-IIIC, with no prior esophageal resection. Neoadjuvant therapy given prior to presentation at MSKCC will be accepted.
* Anticipated to undergo surgical resection (Ivor Lewis, Trans Hiatal, thoracoabdominal, or McKeown procedure) of esophageal cancer either by open or minimally invasive methods
* Chest and abdomen CT scan
* Ability to speak read and write English.

Exclusion Criteria:

* Inability to give informed consent
* Patients requiring a laryngectomy or colon interposition as part of their surgical resection.
* Patients with scleroderma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Thoracic Surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2012-03-14 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

PRIMARY OUTCOMES:
short-term pain | 4 months
  Pain intensity (average of the four pain severity items) measured by BPI at Post-op Days 1 and 3, after epidural removal, at first post-operative clinic visit, at 4 months
short -term quality of life (QOL) | 4 months
  FACT-E score at the post-op visit and at the 4 months

SECONDARY OUTCOMES:
long-term pain | 2 years
  Pain intensity assessed by BPI at 8 months, 12 months, 18 months, 24 months (average of the four pain severity items) Presence of symptoms with intensity ≥3, as assessed by the Symptom Assessment Scale at post-op visit, at 4 months visit (adjusted for pre-operative symptom intensity )
long time quality of life (QOL) | 2 years
  FACT- E score at 8 months, 12 months, 18 months, 24 months. Presence of symptoms with intensity ≥3, assessed by the Symptom Assessment Scale at 8 months, 12 months, 18 months, 24 months
differences in surgical outcomes | 90 days
  operative time, estimated blood loss, length of hospital stay, ICU admission rates, ICU days, complication type, rates and severity as determined by the Common Terminology Criteria for Adverse Events (CTCAE) utilized by MSKCC, rate of anastomotic leak, rate of anastomotic stricture, 90-day (post-operative) hospital readmission rates, time to oral intake, and time to first ambulation.
Complications | 90 days
  operative time, estimated blood loss, length of hospital stay, ICU admission rates, ICU days, complication type, rates and severity as determined by the Common Terminology Criteria for Adverse Events (CTCAE) utilized by MSKCC, rate of anastomotic leak, rate of anastomotic stricture, 90-day (post-operative) hospital readmission rates, time to oral intake, and time to first ambulation.

OTHER OUTCOMES:
predict EUS T3/T4/stricture disease | 2 years
  To evaluate whether a combination of a dysphagia score of 2-4 and a specific CT scan maximal tumor thickness. the patient's CT scan (either performed elsewhere or at MSK) will be reviewed by one radiologist, who will assess the maximal thickness of tumor involvement (>=cm). Patients will then undergo their planned a staging Endoscopic ultrasonography (EUS) by the gastroenterology service, at which time the EUS depth of invasion will be assigned. The dysphagia score and CT thickness will then be compared to the EUS depth (considered the 'gold standard')
predict EUS T3/T4/stricture or earlier EUS disease | 2 years
  the patient's CT scan (either performed elsewhere or at MSK) will be reviewed by one radiologist, who will assess the maximal thickness of tumor involvement (>=cm). Patients will then undergo their planned staging Endoscopic ultrasonography (EUS) by the gastroenterology service, at which time the EUS depth of invasion will be assigned. The dysphagia score and CT thickness will then be compared to the EUS depth (considered the 'gold standard')

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bott, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/